CLINICAL TRIAL: NCT05036993
Title: A Randomized Trial to Investigate the Impact of Professional Development Coaching for MGH Faculty
Brief Title: Investigating the Impact of Professional Development Coaching for Faculty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kerri Palamara McGrath, MD, Director, Center for Physician Well-being, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019P003587
Record Dates: First submitted 2021-08-30; First posted 2021-09-08 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Burnout; Burnout, Professional
Keywords: physician burnout; physician well-being; coaching; faculty development; engagement
MeSH Terms: conditions — Burnout, Psychological; Burnout, Professional

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with crossover to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Coaching
  Interventions: Behavioral: Coaching
- Control (Experimental): Control, Coaching later
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: Coaching — Faculty will be paired with a certified coach who is also a faculty member and receive 6 sessions of coaching over 3 months

SUMMARY:
Coaching is used in business and many other career paths to help the individual define and create their own goals and strategies for achieving those goals. In 2017 the investigators began to investigate the impact of coaching compared to non-coached peers in a randomized trial among non-internal medicine residency programs and internal medicine subspecialty fellowship to understand the impact of this program and its generalizability. Data from all these studies has suggested that coaching is effective in allowing trainees to understand their development over time, find meaning and purpose in their work, and identify their strengths and how to use these to overcome challenges and stressors. Additionally, there is a benefit to the coaches themselves, who can connect with other faculty coaches in a rewarding way, that provides faculty development in leadership development and positive psychology, and space to interact with a group of like-minded physicians.

From the work the investigators have done with housestaff through the MGH Professional Development Coaching Program we have seen a tremendous interest from faculty members for access to similar services. Prior studies show improvement in faculty burnout and engagement at work through small-group sessions focused on reducing distress and promoting well-being. The investigators have also seen that while the training of novice coaches in positive psychology is sufficient to begin crucial conversations about drivers of well-being, the need for more in-depth coaching with certified coaches exists. The goal of this project is to expand coaching to MGH faculty members and provide more in-depth training for coaches through the International Federation of Coaching, through the Wellcoaches Coach Training Program. This is a unique approach to professional development within the field of medicine that has not yet been employed or studied. There was a recent publication of professional coaches hired outside of the field for faculty development, but there has been no training of medical colleagues with professional coaching skills. This has the potential to provide new data for the field and become a sustainable intervention for MGH in addressing ongoing professional development for our faculty and the burnout epidemic. Finally, this can serve as model for implementation in other institutions.

DETAILED DESCRIPTION:
Objectives:

1. Create space for periodic reflection and goal setting for MGPO faculty to visualize their career progress and trajectory.
2. Provide an avenue for MGPO faculty to be trained as professional peer coaches.
3. Maximize the potential for continued professional development for MGPO faculty.
4. Improve burnout, professional fulfillment, resilience, and self-efficacy for MGPO faculty by re-inforcing coping skills and strengths.
5. Evaluate whether professional development coaching by trained faculty peer coaches reduces burnout, improves emotional well-being and improves professional fulfillment in MGPO faculty coaches.

Hypothesis: MGPO Faculty will benefit from a Professional Development Coaching Program in the following ways:

1. A Professional Development Coaching Program, will improve faculty well-being, compared to non-coached controls.
2. A Professional Development Coaching Program will improve faculty workplace satisfaction, compared to non-coached controls.
3. A Professional Development Coaching Program will decrease burnout for faculty participants and faculty coaches and improve their resiliency by allowing them to visualize their accomplish-ments, improve their response to stress of uncertainty, and decrease emotional exhaustion, com-pared to controls.
4. A Professional Development Coaching Program will improve faculty coach well-being, com-pared to non-coach controls.

III. SUBJECT SELECTION

1. Inclusion/exclusion criteria Inclusion criteria for faculty participants to receive coaching: faculty within the Mass General Physicians Organization (MGPO), no specific age range, screening based on self-referral through email Inclusion criteria for faculty participants to become a coach: faculty within the MGPO, no specific age range, screening based on self-referral and information provided in a standard application assessing motivation to become a faculty coach
2. Source of subjects and recruitment methods MGPO Faculty will be sent an email to make them aware of the program for voluntary enrollment. It will be clearly described that their participation is not mandatory.

IV. SUBJECT ENROLLMENT

1. Methods of enrollment, including procedures for patient registration and/or randomization

   MGPO Faculty will be sent an email to make them aware of the program for voluntary enrollment, including both the opportunity to receive coaching in the trial or to become a trained coach. These surveys will serve no evaluative purpose in their job performance. It will be clearly described that their participation is not mandatory. Participants interested in receiving coaching will be placed into 2 groups via simple randomization. Randomization will be carefully done to ensure gender and department other demographics are balanced between the groups. Participants interested in becoming a trained coach will fill out a short application of interest from which 15 individuals will be selected to participate in coach training.
2. Procedures for obtaining informed consent (including timing of consent process) Participants will be invited via email as described above. Details of the study will be included in the email. Electronic consent will be obtained upon declaring interest in the program, as well as in emails when surveys are sent out.
3. Treatment assignment, and randomization (if applicable) Randomization will place participants interested in receiving coaching in 2 groups, either coaching for 3 months, or usual mentoring and well-being practices that exist in their department and through MGH. Randomization will be carefully done to ensure gender and faculty department are balanced between the groups. At the 3 month mark these groups will switch and faculty that were randomized to usual mentoring will be assigned a trained faculty coach for an additional 3 months. Participants will have access to the biographies of trained coaches after being assigned to receive coaching in their respective groups and will be able to select a coach they feel best matches their needs pending coach availability.

V. STUDY PROCEDURES

1. Study visits and parameters to be measured (e.g., laboratory tests, x-rays, and other testing) Participants will be enrolled and followed with data collection for 9 months. 3 months of that time will be spent with a professional development coach with a meeting lasting 30 minutes to 1 hour every 2 weeks. All data collection will be done via survey online at the specified time point. Each coaching session will occur over a secure media platform by Bongomedia. This platform has been adopted by leadership at MGH and will provide deidentified, anonymized contect of the coaching sessions for program leadership. Coaches and participants being coached will have the opportunity to opt out of use of this platform.
2. Drugs to be used (dose, method, schedule of administration, dose modifications, toxicities), include Toxicity Grading Scale (if applicable) N/A
3. Devices to be used N/A
4. Procedures/surgical interventions, etc. N/A
5. Data to be collected and when the data is to be collected Several previously validated survey tools will be utilized for data collection including the Professional Fulfillment Index, the Self Valuation Scale, the Ultrecht Work Engagement Scale, Abbreviated Maslach Burnout Inventory and a Negative Impact of Work on Relationships Scale. Data will be collected at enrollment, 3 months, 6 months and 9 months. All surveys will be filled out by both participants enrolled and randomized for coaching and by trained faculty coaches. These surveys will be sent at enrollment, 3 months, 6 months and 9 months. In addition, both groups will fill out an intervention assessment after sessions that will gather data on themes addressed in the sessions and how effective the sessions felt to the participant. Additionally, all sessions conducted on the Bongomedia platform will produce deidentified, anonymized content that will be aggregated for re-view.

VI. BIOSTATISTICAL ANALYSIS

1. Specific data variables being collected for the study (e.g., data collection sheets).

   Demographic data including gender, number of years as faculty and department will be collected. Survey data will be collected based on scales previously noted.
2. Study endpoints We will survey the faculty with an assessment of the Professional Development Coaching Program at enrollment, 3 months, 6 months and 9 months. After the 9 month survey the study will be completed.
3. Statistical methods Assistance with statistical data analysis will be requested through the Department of Medicine. We will use two-sample t-tests or Wilcoxon rank sum test, whichever more appropriate to compare be-tween groups for the changes from baseline at the different time points for all metrics between the faculty coaches and faculty participants. We will include all subjects in the primary comparisons and explore subgroup analysis stratified by participant characteristics (sex, sub-specialty department)

ELIGIBILITY:
Inclusion Criteria:

* current MGPO Faculty member

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Burnout | 3 months
  Professional Fulfillment Index;Items are scored 0 to 4. Each dimension is treated as a continuous variable. Scale scores are calculated by averaging the item scores of all the items within the corresponding scale. Scale scores can then be multiplied by 25 to create a scale range from 0 to 100. Higher score on the professional fulfillment scale is more favorable. In contrast, higher scores on the work exhaustion or interpersonal disengagement scales are less favorable. Dichotomous burnout categories are determined from the average item score (range 0 to 4) of all 10 burnout items (work exhaustion and interpersonal disengagement), using a cut-point of 1.33. Dichotomous professional flfillment is recommended at an average item score cut-point of >3.0.
Professional Fulfillment | 3 months
  Professional Fulfillment Index; Items are scored 0 to 4. Each dimension is treated as a continuous variable. Scale scores are calculated by averaging the item scores of all the items within the corresponding scale. Scale scores can then be multiplied by 25 to create a scale range from 0 to 100. Higher score on the professional fulfillment scale is more favorable. In contrast, higher scores on the work exhaustion or interpersonal disengagement scales are less favorable. Dichotomous burnout categories are determined from the average item score (range 0 to 4) of all 10 burnout items (work exhaustion and interpersonal disengagement), using a cut-point of 1.33. Dichotomous professional flfillment is recommended at an average item score cut-point of >3.0.
Engagement | 3 months
  Ultrecht Engagement Scale; The UWES utilizes three scales to determine the level of work engagement:
  Vigor, dedication, and absorption. It is a test of how to measure work engagement both on an individual and on group level:Score ranges from 0 to 6 for each item; scores are summed. Higher is better.
Work Relationships | 3 months
  Negative Impact of Work on Relationships; 4 questions with Likert scale 0 to 4, responses summed, higher is worse

SECONDARY OUTCOMES:
Quality of Life Rating | 3 months
  Quality of Life scale - rate quality of life on a scale of 0 to 100, higher is better
Likelihood to leave or reduce | 3 months
  Likelihood to leave or reduce time, report likelihood to leave the institution or reduce clinical time on likert scale 0 to 5; higher is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Palamara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiser SB, Sterns JD, Lai PY, Horick NK, Palamara K. Physician Coaching by Professionally Trained Peers for Burnout and Well-Being: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245645. doi: 10.1001/jamanetworkopen.2024.5645. PMID 38607628